CLINICAL TRIAL: NCT06430489
Title: Treatment of Suicidal Ideation in the Emergency Department Using Nitrous Oxide - PROTORISC Pilote
Brief Title: Treatment of Suicidal Ideation in the Emergency Department Using Nitrous Oxide
Acronym: PROTORISC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR230123
Record Dates: First submitted 2024-04-26; First posted 2024-05-28 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Suicidal Ideation; Emergency Psychiatric; Nitrous Oxide
MeSH Terms: conditions — Suicidal Ideation | interventions — Nitrous Oxide; Air

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical air administration (Placebo Comparator)
  Interventions: Drug: Medical air
- Nitrous oxide administration (Experimental)
  Interventions: Drug: Nitrous oxide

INTERVENTIONS:
Drug: Nitrous oxide — inhaled nitrous oxide (1 hour at 50% concentration)
  Arms: Nitrous oxide administration
Drug: Medical air — inhaled medical air (1 hour)
  Arms: Medical air administration

SUMMARY:
Suicide prevention is a major public health concern, with nearly 9,000 suicides and over 200,000 suicide attempts reported each year in France. Suicide attempts and suicidal ideation are among the most frequent reasons for emergency room visits and psychiatric hospitalizations. Although there is no approved pharmacological treatment for suicidal crises, some psychiatric treatments appear promising. Ketamine, an N-methyl-D-aspartate (NMDA) receptor antagonist, has shown promising results in reducing suicidal ideation. However, its use is limited due to its side effects. Nitrous oxide, another NMDA receptor inhibitor commonly used in anesthesia and pain management, has demonstrated rapid antidepressant effects and few side effects. Given its rapid and lasting effects, nitrous oxide could swiftly alleviate suicidal ideation.

ELIGIBILITY:
Inclusion Criteria:

* Active suicidal ideations
* Beck Scale for Suicidal Ideation score greater than or equal to 8
* French speaking
* Patient admitted to psychiatric emergency department
* Capable of wearing a facial mask
* Having signed an informed consent
* Affiliated with social security

Exclusion Criteria:

* Psychotic disorder, neurodegenerative disease, known substance use disorder (excluding caffeine or tobacco), substance intoxication, unstable somatic pathology
* Pregnancy or breastfeeding
* Contraindication to the use of nitrous oxide
* Legal incapacity
* Participation in another drug clinical trial
* Patient subject to compulsory care measures

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
suicidal ideation severity | At Hour 4
  Suicidal ideation severity decrease (SSI)

SECONDARY OUTCOMES:
suicidal ideation severity | At Hour 24, at Hour 48, at Day 7 and at Month 1
  Suicidal ideation severity decrease (SSI): The score ranges from 0 to 38. The higher the total score, the greater the severity of suicide ideation
Suicidal ideation assessed by the SSI scale. | At Hour 24, at Hour 48, at Day 7 and at Month 1
Suicidal ideation assessed by the Columbia Suicidal Risk Severity Scale (C-SSRS). | At Day 0 and Day 7
Depressive symptoms measured by hetero-assessment using the "Montgomery-Asberg Depression Rating Scale" (MADRS). | At Day 0 and Day 7
  The higher the total score, the greater the severity of depression
Depressive symptoms measured by the "Patient Health Questionnaire" PHQ-9 self-administered questionnaire. | At Day 0, At Hour 4, at Hour 24, at Hour 48 and at Day 7
  The higher the total score, the greater the severity of depression
Intensity of anxiety measured by the "State and Trait Anxiety Inventory" (STAI) scale. | At Day 0 up to Hour 4, at Hour 24, at Hour 48 and at Day 7
  The higher the total score, the greater the severity of anxiety
Overall improvement measured by change in Clinical Global Impression - Improvement (CGI) scale score. | At Day 0 up to Hour 4, at Hour 24, at Hour 48 and at Day 7
  The higher the score, the more the clinical condition has worsened
Commitment to suicidal action in the month following inclusion | in the month following Day 0
  Number of suicide attempts and methods in the month following the intervention
Consumption of psychotropic medication for anxiolytic or sedative purposes. | At Hour 0 up to Hour 4

CONTACTS AND LOCATIONS:
Overall Officials: ANAIS VANDEVELDE, MD, PHD, Principal Investigator — CHRU de Tours
Locations (1):
- Psychiatric Emergencies, Tours, France

IPD SHARING:
Plan to Share IPD: No